CLINICAL TRIAL: NCT05250713
Title: Quantification of the Immediate Impact of Weak Electric Fields on Brain Activity by SEEG Measurements in Drug-resistant Focal Epilepsy Patients
Brief Title: Evaluation of Direct Effects of Electric Fields on Brain
Acronym: GALVANI PS-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2020-66; ID-RCB (Other: 2021-A00529-32)
Record Dates: First submitted 2022-01-30; First posted 2022-02-22 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Epilepsy
Keywords: tDCS (transcranial direct current stimulation); tACS (transcranial alternate current stimulation); Starstim; transcranial stimulation; SEEG (stereoelectroencephalography)
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (Experimental): Patients receiving tDCS during SEEG investigation
  Interventions: Device: Transcranial stimulation
- tACS (Experimental): Patients receiving tACS during SEEG intervention
  Interventions: Device: Transcranial stimulation

INTERVENTIONS:
Device: Transcranial stimulation — Patients will receive either direct current stimulation or alternate stimulation.

SUMMARY:
Transcranial current stimulation (tCS), a safe, tolerable technique employing weak currents (~ 1 mA) applied to the scalp, has been shown to be a promising technique in alleviating seizures in focal epilepsy patients. Although studies reveal a decrease in the epileptiform activity due to tCS, this field lacks a quantification of neurophysiological changes during and immediately after stimulation. The investigators hypothesise that tCS can effectively reduce the amplitude and rate of interictal spikes as well as the functional connectivity between regions during and immediately after stimulation. It is thus planned to deliver an extensive quantitative description of the tCS effects on interictal spike activity, functional connectivity and other tissue biomarkers, using the simultaneous recording of intracranial signals during tCS. Moreover, the investigators seek to compare these variations between different tCS paradigms (direct current -tDCS- vs alternate current -tACS- stimulation).

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Male or female, aged ≥ 18 years old
3. Focal drug-resistant epilepsy
4. Patient undergoing a clinical SEEG investigation
5. Stated willingness to comply with all study procedures and availability for the duration of the study
6. Patient affiliated or beneficiary of a health insurance plan
7. Patient for whom MRI images (3D T1) are exploitable and fit with the minimum MRI requirements needed for biophysical modelling (cf annex in 14.), prior to SEEG electrodes implantation
8. Patient for whom a CT-scan with electrodes (or MRI with electrodes) has been realized after SEEG procedure.

Exclusion Criteria:

1. Difficulty to read or understand the French language, or inability to understand the information regarding the study
2. Person protected by articles L1121-5, L1121-6 and L1121-8 of Public Health Code (pregnant or breastfeeding woman, deprived of liberty by judicial decision, situations of social fragility, adults or unable to express their consent). Pregnancy will be evaluated during screening with a urine pregnancy test.
3. Presence of severe negative outcome of SEEG surgery preventing the acquisition of SEEG data (i.e. hemorragic complications, subcutaneous infection), at the time of inclusion.
4. Patient showing contraindications for electric stimulation at the time of inclusion:

   (A) Patient with unstable or non-controlled neuropsychiatric illness (B) Patients having cardiac or medication implants (C) Patients with implanted pacemakers (D) Patients with serious brain injury (E) Patients showing damage of skin at sites of stimulation
5. Any condition that, according to the investigator, is not compatible with carrying out the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-04-26 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Measure of epileptogenic markers in intracranial brain signals recordings | During tDCS or tACS
  Rate and amplitude of interictal epileptogenic spikes
Measure of epileptogenic markers in intracranial brain signals recordings | After tDCS or tACS
  Rate and amplitude of interictal epileptogenic spikes
Measure of functional connectivity in intracranial brain signals recordings | During tDCS or tACS
  Neural network excitability
Measure of functional connectivity in intracranial brain signals recordings | After tDCS or tACS
  Neural network excitability

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — AP-HM
Locations (1):
- Service Epileptologie et Rythmologie Cérébrale, Marseille, France

IPD SHARING:
Plan to Share IPD: No